CLINICAL TRIAL: NCT02055521
Title: Search Tolerance Signature in Vascularised Composite Allograft
Acronym: BIOCTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: ISTITUTO ITALIANO CHIRURGIA DELLA MANO, Italy (Unknown); medizinische universität innsbruck, Austria (Unknown); Hospital Clínico Universitario de Valencia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013.815
Record Dates: First submitted 2014-01-17; First posted 2014-02-05 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Hand and Face Allotransplantation
Keywords: Composite tissue allograft; operational tolerance; skin rejection; Hand and Face allotransplantation
MeSH Terms: interventions — Blood Specimen Collection; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood sample, biopsy

SUMMARY:
Composite tissue allotransplants (CTA) involve transplantation of various tissues including vessels, nerves, skin, bones, and immune cells and entail a significant antigenic load. The large majority of recipients have been maintained on immunosuppression therapy similar to that used in solid organ transplantation that is associated with the complications usually reported in solid organ transplantation. The question whether risks associated with indefinite immunosuppressive are justified for a non-lifesaving procedure still remains unanswered. At present no CTA recipient proved to be spontaneously tolerant with any immunosuppressive protocol; indeed, until now all recipients who discontinued the immunosuppressive therapy rejected their graft. On the other hand CTA recipients showed a low incidence of chronic rejection despite the high incidence of acute rejection episodes.

For all these reasons it should be of great interest to minimize the immunosuppression in CTA patients knowing their immunologic "risk". The main outcome of this study is to search for the signature of tolerance in recipients of hand or face allotransplantation testing biomarkers previously identified in operational tolerant kidney transplant recipients.

These markers have been developed studying tolerant kidney recipients and they were already tested in five bilateral hand transplantations and one face transplantation.

The present study will include hand and face allograft recipients transplanted at least one year in several European institutions (Innsbruck, Lyon, Monza, Valencia): 11 bilateral hand transplantations, 4 single hand transplantations and 3 face transplantations. All the patients will undergo B cell phenotyping, TCR repertoire, molecular signature from operational tolerance and a skin biopsy with immunohistochemical staining of the specimens in order to show signs of acute or chronic rejection.

The results could provide a valid tool to detect operationally tolerant recipients as well as recipients prone to develop chronic rejection.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Hand (unilateral/bilateral) or face allotransplantation for at least one year
* Patient without clinical sign of acute rejection at inclusion
* Patient who signed the informed protocol consent
* Patient older than 18 years old
* Patient covered by an health insurance
* Patient without legal protection

Exclusion Criteria:

* Patient with Hand or face allotransplantation for less than one year
* Patient with clinical sign of acute rejection at inclusion
* Unsigned protocol consent
* Patient under the age of 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Biomarkers of molecular signature from operational tolerance and/or chronic rejection research | 1 day
  B cell phenotyping, TCR repertoire, molecular signature from operational tolerance

SECONDARY OUTCOMES:
Pathological characteristics of skin acute/chronic rejection on skin biopsy | 1 day
  skin biopsy with immunohistochemical staining of the specimens in order to show signs of acute or chronic rejection. We will try to correlate the signature of tolerance with the absence of chronic rejection symptoms, both clinically and in skin protocol biopsies.
Phenotype of skin T lymphocyte in cutaneous biopsies | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Background] Emmanuel Morelon, Sophie BROUARD, Stephan Schneeberger, Anne-Marie Weissenbache. Abstract accepted for presentation at the IHCTAs Congress (Philadelphia, April 2015) and at the ESOT Congress (Brussels, September 2015)."